CLINICAL TRIAL: NCT00103207
Title: Phase II Study of C225 (Cetuximab) for the Treatment of Patients With Advanced Bronchioalveolar Carcinoma (BAC) or Adenocarcinoma With BAC Features
Brief Title: Cetuximab in Treating Patients With Recurrent or Stage IIIB or Stage IV Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000409755; U10CA021115 (NIH); E1504 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: bronchioalveolar carcinoma (BAC); adenocarcinoma with BAC features; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; cetuximab
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab (Experimental): Cetuximab was given as a weekly intravenous (IV) infusion (over 60 minutes) at 250 mg/m2 from week 2 onwards after an initial loading dose of 400 mg/m2 (over 120 minutes) on week 1 until disease progression or unacceptable toxicity. The infusion rate of cetuximab could not exceed 5 mL/min. Each cycle will be 28 days in length. To prevent a hypersensitivity reaction, all patients were premedicated with diphenhydramine hydrochloride 50 mg (or an equivalent antihistamine) by IV (over 30-60 minutes) prior to the first dose of cetuximab. Premedication might be administered prior to subsequent doses, but at the investigator's discretion, the dose of diphenhydramine (or a similar agent) was reduced.
  Interventions: Biological: cetuximab

INTERVENTIONS:
Biological: cetuximab
  Other Names: C225

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well cetuximab works in treating patients with recurrent or stage IIIB or stage IV lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with recurrent or stage IIIB or IV bronchoalveolar carcinoma (BAC) or adenocarcinoma of the lung with BAC features treated with cetuximab.

Secondary

* Determine the overall survival and time to progression in patients treated with this drug.
* Determine the toxic effects of this drug in these patients.
* Correlate expression of total and phosphorylated epidermal growth factor receptor (EGFR), total and phosphorylated AKT3, and total and phosphorylated MAPKinase with response in patients treated with this drug.
* Determine whether the presence of polymorphisms or mutations in the EGFR gene influences response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1-2 hours once on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ACTUAL ACCRUAL: A total of 72 patients were accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically or cytologically confirmed bronchoalveolar carcinoma (BAC) or adenocarcinoma of the lung with BAC features meeting 1 of the following stage criteria:

  * Stage IIIB disease (with pleural or pericardial effusion)
  * Stage IV disease
  * Recurrent disease
* Measurable disease
* Tumor tissue available from biopsy
* Age of 18 and over
* ECOG performance status of 0-2
* Life expectancy greater than 3 months
* White blood cell (WBC) ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* Aspartate aminotransferase (AST) and/or alanine aminotranferease (ALT) ≤ 2.5 times upper limit of normal
* Creatinine normal OR Creatinine clearance ≥ 60 mL/min
* No more than 1 prior chemotherapy regimen for advanced BAC
* More than 3 years since prior chemotherapy for other malignancies
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) for this malignancy and recovered
* HIV-positive patients are eligible provided the following criteria are met:

  * CD4 count ≥ 100/mm^3
  * Undetectable viral load within the past 3 months
  * Receiving a stable antiretroviral regimen for ≥ 4 weeks before study entry
* Fertile patients must use effective contraception
* At least 2 weeks since prior radiotherapy and recovered

EXCLUSION CRITERIA:

* Untreated brain metastases

  * Patients with stable brain metastases ≥ 4 weeks after external beam radiotherapy to the brain are eligible
* Acute hepatitis
* Symptomatic congestive heart failure
* Uncontrolled hypertension
* Unstable angina pectoris
* Cardiac arrhythmia
* Pregnant or nursing
* Prior allergic reaction to chimerized or murine monoclonal antibody therapy
* Documented presence of human anti-mouse antibodies
* Ongoing or active infection
* Psychiatric illness or social situation that would preclude study compliance
* Other uncontrolled illness
* Prior cetuximab
* Concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)
* Other prior known epidermal growth factor receptor inhibitors (e.g., gefitinib or erlotinib)
* Other concurrent investigational agents
* Other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-10-13 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, MD, Study Chair — Emory Winship Cancer Institute
Locations (157):
- United States (157):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Morton Hospital & Medical Center, Taunton, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Result] Ramalingam SS, Lee JW, Belani CP, Aisner SC, Kolesar J, Howe C, Velasco MR, Schiller JH. Cetuximab for the treatment of advanced bronchioloalveolar carcinoma (BAC): an Eastern Cooperative Oncology Group phase II study (ECOG 1504). J Clin Oncol. 2011 May 1;29(13):1709-14. doi: 10.1200/JCO.2010.33.4094. Epub 2011 Mar 21. PMID 21422434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on August 10, 2005, accrued its first patient on October 13, 2005, and closed to accrual on December 12, 2008 with final accrual of 72 patients.
Groups:
- Cetuximab: Cetuximab was given as a weekly intravenous (IV) infusion (over 60 minutes) at 250 mg/m2 from week 2 onwards after an initial loading dose of 400 mg/m2 (over 120 minutes) on week 1 until disease progression or unacceptable toxicity. The infusion rate of cetuximab could not exceed 5 mL/min. Each cycle will be 28 days in length. To prevent a hypersensitivity reaction, all patients were premedicated with diphenhydramine hydrochloride 50 mg (or an equivalent antihistamine) by IV (over 30-60 minutes) prior to the first dose of cetuximab. Premedication might be administered prior to subsequent doses, but at the investigator's discretion, the dose of diphenhydramine (or a similar agent) was reduced.
  Only eligible patients with confirmed diagnosis are included in the main analysis.
Period: Overall Study
Arm/Group | Cetuximab
Started | 72
Eligible Patients w/ Confirmed Diagnosis | 41
Eligible Patients w/ Smoking Status Data | 37
Completed | 34
Not Completed | 38
Not completed — Adverse Event | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Other complicating disease | 1
Not completed — Ineligible | 4
Not completed — Diagnosis of BAC not confirmed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 70 [26 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Proportion of Patients With Objective Response)
Description: Response was evaluated using RECIST 1.0 criteria. Per RECIST criteria, Complete response (CR)= disappearance of all target and nontarget lesions Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits. Objective response = CR + PR.
Time Frame: Assessed every 8 weeks during treatment; after off-treatment, every 3 months for 2 years and then every 6 months for 3 years
Population: Only eligible and treated patients with confirmed diagnosis are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion
Arm/Group | Cetuximab
Number analyzed (Participants) | 41
Proportion | 0.07 [0.02 to 0.18]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from registration to death.
Time Frame: Every week during treatment; after off-treatment, every 3 months for 2 years and then every 6 months for 3 years
Population: Only eligible and treated patients with confirmed diagnosis are included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab
Number analyzed (Participants) | 41
Months | 17.9 [10.6 to 31.5]

3. Secondary Outcome: Time to Progression
Description: Time to progression is defined as time from study entry until disease progression. Progression is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s) or unequivocal progression of existing nontarget lesions.
Time Frame: as for outcome 1
Population: Only eligible and treated patients with confirmed diagnosis are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab
Number analyzed (Participants) | 41
Months | 3.8 [2.6 to 5.7]

4. Secondary Outcome: Overall Survival by Smoking Status
Description: Medians of overall survival by smoking status are reported.
Time Frame: Overall survival assessed every week during treatment; after off-treatment, every 3 months for 2 years and then every 6 months for 3 years. Smoking status evaluated at baseline
Population: Only eligible and treated patients with confirmed diagnosis and smoking status data are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Never Smoker: Eligible and treated patients who never smoked.
- Former/Current Smoker: Eligible and treated patients who are former or current smokers.
Arm/Group | Never Smoker | Former/Current Smoker
Number analyzed (Participants) | 7 | 30
Months | 40.9 [7.2 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 15.5 [8.9 to 30.2]

5. Secondary Outcome: Time to Progression by Smoking Status
Description: Medians of time to progression by smoking status are reported.
Time Frame: Progression assessed every 8 weeks during treatment; after off-treatment, every 3 months for 2 years and then every 6 months for 3 years. Smoking status evaluated at baseline
Population: Only eligible and treated patients with confirmed diagnosis and smoking status data are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Never Smoker | Former/Current Smoker
Number analyzed (Participants) | 7 | 30
Months | 2.6 [1.8 to 6.0] | 3.7 [2.6 to 5.7]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment.
Groups:
- Cetuximab: All treated patients were evaluated for toxicities.
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 27/72
Other Adverse Events (participants affected / at risk) | 70/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=72)
Allergic reaction (Immune system disorders) | 1
Lymphopenia (Investigations) | 1
Fatigue (General disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 2
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 11
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, ungual (Infections and infestations) | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1
Creatinine, increased (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Head/headache (Nervous system disorders) | 1
Skin, pain (Skin and subcutaneous tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=72)
Allergic reaction (Immune system disorders) | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Anemia (Blood and lymphatic system disorders) | 27
Leukocytes, decreased (Investigations) | 8
Neutrophils, decreased (Investigations) | 7
Platelets, decreased (Investigations) | 5
Fatigue (General disorders) | 44
Fever w/o neutropenia (General disorders) | 8
Rigors/chills (General disorders) | 4
Weight loss (Investigations) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 19
Nail changes (Skin and subcutaneous tissue disorders) | 10
Pruritus/itching (Skin and subcutaneous tissue disorders) | 14
Rash/desquamation (Skin and subcutaneous tissue disorders) | 22
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 60
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 9
Skin-other (Skin and subcutaneous tissue disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 15
Constipation (Gastrointestinal disorders) | 16
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 22
Dyspepsia (Gastrointestinal disorders) | 4
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 6
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 23
Taste disturbance (Nervous system disorders) | 9
Vomiting (Gastrointestinal disorders) | 8
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5
Edema limb (General disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Alkaline phosphatase increased (Investigations) | 8
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4
Creatinine, increased (Investigations) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 32
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 20
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 6
Dizziness (Nervous system disorders) | 4
Neuropathy-sensory (Nervous system disorders) | 6
Dry eye syndrome (Eye disorders) | 4
Head/headache (Nervous system disorders) | 11
Muscle, pain (Musculoskeletal and connective tissue disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No